CLINICAL TRIAL: NCT03692572
Title: Influence of Early Menopause on Sympathetic Activation and Cardiovascular Function in Older Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Texas Health Resource (Unknown)
Responsible Party: Principal Investigator, Qi Fu, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: STU 032018-052
Record Dates: First submitted 2018-09-25; First posted 2018-10-02 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Early Menopause; Menopause
Keywords: Neural control; Cardiovascular function; Inorganic nitrate supplementation
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Intervention Model Description: 2 groups of women (early and normal menopause transition) will be enrolled to crossover design study in a fashion of randomized and double-blinded.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only research nurse will have an access to the randomization sheet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate supplementation (Active Comparator): Nitrate rich (6.8 mmol) beet root juice (70ml) twice a day
  Interventions: Dietary Supplement: Nitrate supplementation
- Placebo (Placebo Comparator): Nitrate depleted (0.04 mmol) placebo juice (70ml) twice a day
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Nitrate supplementation — Subjects will drink 70 ml of beet root juice twice a day for 2 weeks.
  Arms: Nitrate supplementation
Dietary Supplement: placebo — Subjects will drink 70 ml of nitrate depleted placebo juice twice a day for 2 weeks.
  Arms: Placebo

SUMMARY:
Women who enter menopause early are at a greater risk for developing cardiovascular disease later in life as compared to women with normal onset of menopause. This increased risk may be due to a prolonged length of time with decreased hormone levels post-menopause; however, this health risk remains understudied. The current study plan to study why women with early menopause are at higher risk for cardiovascular disease by evaluating their sympathetic nervous system and heart-blood vessel function. In addition, there is lack of promising treatment plans for cardiovascular disease in post-menopausal women. Therefore, the current study will also test the impact of dietary nitrate on post-menopausal women to determine if it might serve as a potential treatment to reduce risk of cardiovascular disease in older women.

DETAILED DESCRIPTION:
The current study is recruiting two groups of women aged between 60-70 years old; 1) women who had early natural/non-surgical menopause (age 40-44 yrs) and 2) women who had normal natural/non-surgical menopause (age 50-54). The investigators are recruiting women who do not have any cardiovascular disease, hypertension, diabetes, and other major health issue.

The main hypothesis of the project is that early menopause negatively impacts the heart, blood vessel and nerve system due to the increased length of time with reduced hormone levels; which could explain the relationship between early menopause and greater risk of cardiovascular disease in later life. Sympathetic nerve system and cardiovascular functions will be evaluated in both groups to compare the impact of prolonged hormone deficiency. In addition, current study will examine the impact of inorganic nitrate supplementation (beet root juice) to see if there are any favorable changes after 2 weeks of beet root juice intake. There are 2 main test visits in the current study.

Visit 1. Nerve system test (maximally take about 5 hours): Participants will rest in the supine position for ≥ 20 mins. Resting heart rate, breathing rate, finger blood pressure will be monitored. Cardiac output will be assessed using the acetylene gas rebreathing technique (1 hour). IV will be inserted for blood draw. Nerve signal search will be performed using a thin needle behind knee to find a signal from a specific nerve. At the same time, transcranial Doppler probe will be placed on the head to look at brain blood flow using soft head gear (1-2 hour). After acceptable signals are obtained, baseline data collection will begin. It will be followed by handgrip exercise and hand immersion to cold water to examine neural sympathetic response to different stimuli (30 mins). After this, to evaluate nerve response to different degrees of passive standings, a bed will be tilted to 30° and 60° for 8 mins each. Blood samples will be obtained in the supine resting position and at the end of 60° tilt (45 mins).

Visit 2. Heart and vessel function assessment (Proximately take 2 hours): All measurements are non-invasive for this visit. Participants will rest in the supine position for ≥ 20 mins. Resting heart function will be assessed by ultrasound echocardiography (30mins). Vascular stiffness measurement will be performed using a probe placed on wrist, neck and leg groin area (30 mins). Vascular endothelial function will be measured using flow-mediated dilation and followed by smooth muscle responsiveness test will be performed by measuring brachial artery diameter changes for 10 min following 0.4 mg sublingual nitroglycerin administration (1 hour).

After Visit 1-2, participant will be asked to drink either dietary nitrate supplementation or placebo for 2 weeks (randomly assigned). After 2 weeks intervention, participant will come back for post-intervention tests which are identical to visit 1 and 2.

After completion of the first intervention, participants will have at least 2 weeks of wash-out period. After 2 weeks participant will be back to the lab and repeat the visit 1 and 2, as well as 2 weeks of dietary nitrate supplementation or placebo. (For those who received 2 weeks of nitrate supplementation for the first intervention, it will be a placebo for this intervention. For those who received placebo for the first intervention, it will be a nitrate supplementation for this intervention). After intervention participants will repeat the visit 1 and 2 again.

ELIGIBILITY:
Inclusion Criteria:

* Healthy normotensive postmenopausal women
* Current age between 60 and 70 years
* Who have experienced "natural" or non-surgical menopause

Exclusion Criteria:

* Any evidence of cardiopulmonary disease
* History of hormone replacement therapy in the last 5 years
* Chronic kidney disease
* Diabetes mellitus
* Hypertension
* Current abuse of alcohol or drugs and use of tobacco products
* Surgical procedure induced menopause

Ages: 60 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 22 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Muscle sympathetic nerve activity (MSNA) | Change from baseline resting MSNA to 2 weeks post nitrate supplementation resting MSNA
  Muscle sympathetic nerve activity will be measured using microneurography at the peroneal nerve.

SECONDARY OUTCOMES:
Cardiac Echocardiogram | Change from baseline cardiac function to 2 weeks post nitrate supplementation resting cardiac function
  Systolic and diastolic cardiac function will be measured using high resolution ultrasound echocardiogram
Vascular endothelial function | Change from baseline brachial artery endothelial function to 2 weeks post nitrate supplementation brachial artery endothelial function
  Brachial artery endothelial function will be measured using flow-mediated dilation
Arterial stiffness/wave properties | Change from baseline pulse wave velocity and wave reflection to 2 weeks post nitrate supplementation resting pulse wave velocity and wave reflection
  Central and peripheral pulse wave velocity and wave reflection will be assessed using arterial tonometry

CONTACTS AND LOCATIONS:
Overall Officials: Qi Fu, Ph.D., Study Director — Faculty
Locations (1):
- Institute for Exercise and Environmental Medicine, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided